CLINICAL TRIAL: NCT07074717
Title: Penile Skin Versus Buccal Mucosal Graft in Augmentation Urethroplasty for Long Anterior Urethral Stricture: A Prospective Randomized Study
Brief Title: Penile Skin Versus Buccal Mucosal Graft in Augmentation Urethroplasty for Long Anterior Urethral Stricture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ahmed Elmaadawy, Lecturer of Urology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR1074/1/25
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Penile Skin; Buccal Mucosal Graft; Augmentation; Urethroplasty; Long Anterior; Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buccal Mucosal Graft (BMG) (Experimental): Participants will undergo dorsal onlay augmentation urethroplasty using a buccal mucosal graft harvested from the inner cheek. The procedure is performed under spinal or general anesthesia. Graft is sutured dorsally over the strictured urethral segment after excision of the fibrotic tissue.
  Interventions: Procedure: Buccal Mucosal Graft (BMG) Urethroplasty
- Penile Skin Graft (PSG) (Experimental): Participants will undergo dorsal onlay augmentation urethroplasty using a penile skin graft harvested from the ventral surface of the penis. The hairless skin is prepared and sutured dorsally over the strictured urethral segment. The procedure is done under spinal or general anesthesia.
  Interventions: Procedure: Penile Skin Graft (PSG) Urethroplasty

INTERVENTIONS:
Procedure: Buccal Mucosal Graft (BMG) Urethroplasty — Urethroplasty using a buccal mucosal graft harvested from the inner cheek. The graft is dorsally onlaid to reconstruct the strictured urethral segment. The procedure is conducted under spinal or general anesthesia.
  Other Names: Dorsal onlay buccal mucosal graft
  Arms: Buccal Mucosal Graft (BMG)
Procedure: Penile Skin Graft (PSG) Urethroplasty — Urethroplasty using a penile skin graft harvested from the ventral surface of the penis. The graft is applied dorsally after excision of the fibrotic urethral segment. The surgery is performed under spinal or general anesthesia.
  Other Names: Dorsal onlay penile skin graft
  Arms: Penile Skin Graft (PSG)

SUMMARY:
The aim of this study is to analyze the outcomes of dorsal onlay buccal mucosal graft (BMG) and penile skin graft (PSG) urethroplasty in the management of long segment bulbar urethral stricture.

DETAILED DESCRIPTION:
Penile urethral reconstruction proves to be a continuous challenge as no perfect technique is considered for all patients with this problem. Among all the methods used for treatment of urethral stricture, the substitution urethroplasty with tissue transfer using either flap or graft is the gold standard treatment option for long segment urethral strictures.

In 1993, McAninch described a circular fasciocutaneous flap for the management of penile urethral stricture up to 15 cm that showed excellent cosmetic and functional outcomes due to this being a hairless, flexible flap with a rich vascular supply.

Buccal mucosal graft (BMG) was rediscovered and popularized in 1992 by Burger et al., then El-Kassaby et al. in 1993 published a series using buccal mucosal graft to repair anterior urethral stricture. Buccal mucosal graft became an ideal urethral substitute due to easy harvesting, hairlessness and compatibility in a wet environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with long segment anterior urethral stricture that was defined as a stricture with a length of more than 1 cm with spongiofibrosis.
* Patients with previous failed urethral dilatation or direct vision internal urethrotomy (DVIU)

Exclusion Criteria:

* Patients with lichen sclerosus
* Patients with history of hypospadias repair
* Patients with recurrent urethral stricture after failed previous urethroplasty

Min Age: 18 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Success Rate | 9 months postoperatively
  Success is defined as satisfactory urinary stream with no need for further intervention (such as dilatation or DVIU) and no evidence of stricture on retrograde urethrogram during follow-up.

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 9 months postoperatively
  Evaluation of changes in urinary symptoms using International Prostate Symptom Score (IPSS) to assess functional outcome and patient comfort after urethroplasty will be assessed.
Length of Urethral Stricture | Intraoperatively
  Length of Urethral Stricture will be measured to compare the characteristics of strictures managed by each graft technique.
Postoperative Complications | 9 months postoperatively
  Complications such as infection, bleeding, graft failure, and fistula formation following surgery will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia Governorate, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.